CLINICAL TRIAL: NCT02770391
Title: The Association Between HSD3B1 Genotype and Steroid Metabolism in Normal and Prostate Cancer Tissue of Men With Intermediate and High-risk Prostate Cancer Undergoing Radical Prostatectomy After Treatment With Apalutamide and Leuprolide
Brief Title: Apalutamide and Leuprolide in Intermediate and High-risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Moshe Ornstein, MD, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5815
Record Dates: First submitted 2016-05-05; First posted 2016-05-12 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: HSD3B1 Genotype; Steroid Metabolism; High-risk Prostate Cancer; Apalutamide; ARN-509
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apalutamide + Leuprolide Acetate (Experimental): All participating patients will receive a single dose of leuprolide 7.5 mg intramuscularly (IM) in addition to Apalutamide 240 mg orally daily for four weeks prior to radical prostatectomy (RP). Treatment will be started on day (-28) ± 3 from the scheduled RP date to minimize the variability of treatment duration. Apalutamide may be continued up to and including the day before
  Interventions: Drug: Leuprolide acetate; Drug: Apalutamide; Procedure: Radical prostatectomy

INTERVENTIONS:
Drug: Leuprolide acetate — Leuprolide acetate, Intramuscular injection - 7.5 mg, one time dose on day (-28) ± 3
  Other Names: Lupron
Drug: Apalutamide — Apalutamide, PO, 240 mg daily, starting day (-28) ± 3 until the day before radical prostatectomy. Apalutamide will be initiated the same day patients receive their leuprolide acetate injection.
  Other Names: ARN-509
Procedure: Radical prostatectomy

SUMMARY:
This is a research study to test an investigational drug (Not FDA approved), Apalutamide given in combination with Leuprolide acetate (FDA approved) in men diagnosed with high-risk prostate cancer who have already selected to have surgery to remove their prostate gland as part of their treatment plan. The main purpose of this study is to determine how tumors make androgens (male hormones), which makes these tumors more aggressive and resistant to hormonal therapy and how a short period of treatment with Apalutamide and leuprolide acetate prior to surgery can affect the production of these hormones in normal and malignant prostate tissue.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the differential effect of neo-adjuvant leuprolide and Apalutamide on dihydrotestosterone (DHT) concentration in benign prostate tissue based on HSD3B1 genotype.

Secondary Objective(s): To evaluate the differential effect of neoadjuvant leuprolide and Apalutamide on other androgen (testosterone (T), dehydroepiandrosterone (DHEA), androstenediol, 5α-androstanedione (5α-dione), androstenedione (AD), androsterone and 5α-androstanediol) concentrations in benign and malignant prostate tissue based on HSD3B1 genotype.

To compare the level of DHT, T, DHEA, androstenediol, 5α-dione, AD, androsterone and 5α-androstanediol between normal and malignant prostate tissue after neoadjuvant treatment with leuprolide and Apalutamide

To determine the safety of the combination of Leuprolide and Apalutamide administered prior to radical prostatectomy

To evaluate prostatic specific antigen (PSA), FKBP5, TMPRSS2, EZH2, H3K27 and UBE2C tissue expression (via immunohistochemistry (IHC) and quantitative polymerase chain reaction (qPCR)) in benign and malignant prostate tissue after treatment with Leuprolide and Apalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate with histological or cytological confirmation without neuroendocrine differentiation or small cell histology and with G 4+3 or higher, and PSA ≥ 10, and ≥T2b, for whom radical prostatectomy has been recommended and who choose to undergo radical prostatectomy.
* A minimum tissue requirement of ≥3 core biopsies with tumor involvement and at least 50% tumor involvement in one of the core biopsies is required.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hemoglobin of ≥ 10 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count of ≥ 100k/mL independent of transfusion and/or growth factors within 3 months prior to randomization
* Serum albumin ≥3.0 g/dL
* Serum creatinine < 2.0 times the upper limit of normal (ULN) {or a calculated creatinine clearance ≥ 60 mL/min}
* Serum potassium ≥3.5 mmol/L
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN
* Total serum bilirubin levels < 1.5 x ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
* Be capable of swallowing study agents whole as a tablet
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study.
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry.
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

* The use of any prior hormones including luteinizing hormone-releasing hormone (LHRH) agonists , LHRH antagonists, antiandrogens such as bicalutamide, flutamide and nilutamide, and/or the use of 5-alpha reductase inhibitors, prostate cancer (PC) Spes (or PC-x product), Megestrol Acetate, or estrogen containing nutriceuticals within 6 months of study treatment initiation.
* Prior radiation therapy, immunotherapy, chemotherapy or other investigational therapy given for prostate cancer.
* "Currently active" second malignancy other than non-melanoma skin cancers or non-muscle invasive transitional cell carcinoma of bladder. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered (by their physician) to be at less than 30% risk for relapse.
* History of seizure or condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Current systemic steroid therapy (inhaled or topical steroids are also not allowed)
* Have received treatment with any form of therapy with CYP17 inhibitory activity such as ketoconazole, aminoglutethimide, or an antiandrogen such as bicalutamide within 6 months of study treatment initiation.
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids within 6 months of enrollment
* Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
* Have uncontrolled hypertension;subjects with a history of hypertension are permitted in the study provided their blood pressure is controlled by anti-hypertensive therapy, at the discretion of the treating physician
* Have a known history of pituitary or adrenal dysfunction
* Have clinically significant heart disease as evidenced by severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Have a history of gastric bypass surgery or severe malabsorption that may interfere with the absorption of the study agents
* Be taking or require the use of prohibited medications as listed
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ornstein, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Apalutamide + Leuprolide Acetate: All participating patients will receive a single dose of leuprolide 7.5 mg intramuscularly (IM) in addition to Apalutamide 240 mg orally daily for four weeks prior to radical prostatectomy (RP). Treatment will be started on day (-28) ± 3 from the scheduled RP date to minimize the variability of treatment duration. Apalutamide may be continued up to and including the day before
  Leuprolide acetate: Leuprolide acetate, Intramuscular injection - 7.5 mg, one time dose on day (-28) ± 3
  Apalutamide: Apalutamide, PO, 240 mg daily, starting day (-28) ± 3 until the day before radical prostatectomy. Apalutamide will be initiated the same day patients receive their leuprolide acetate injection.
  Radical prostatectomy
Period: Overall Study
Arm/Group | Apalutamide + Leuprolide Acetate
Started | 54
Completed | 48
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Surgery delayed unevaluable | 2
Not completed — Treatment discontinued due to treatment inturruption | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 46
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Dihydrotestosterone (DHT) Concentration in Benign Prostate Tissue After a Combination Drug Treatment Based on Genotype Status
Description: To evaluate the differential effect of neo-adjuvant leuprolide and ARN-509 on dihydrotestosterone (DHT) concentration in benign prostate tissue based on HSD3B1 genotype.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue each gave two samples
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 15
Number analyzed (Tissue Sample) | 30
nM
  homozygous (1245A): number analyzed (Participants) | 8
  homozygous (1245A): number analyzed (Tissue Sample) | 16
  homozygous (1245A) | 9.066 (7.775)
  heterozygous (1254C): number analyzed (Participants) | 5
  heterozygous (1254C): number analyzed (Tissue Sample) | 10
  heterozygous (1254C) | 5.917 (3.458)
  homozygous (1245C): number analyzed (Participants) | 2
  homozygous (1245C): number analyzed (Tissue Sample) | 4
  homozygous (1245C) | 9.345 (5.607)

2. Secondary Outcome: Other Androgens Concentration in Benign Prostate Tissue After Neo-adjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate the differential effect of neoadjuvant leuprolide and ARN-509 on other androgens (testosterone (T), dehydroepiandrosterone (DHEA), androstenediol, 5?-androstanedione (5?-dione), androstenedione (AD), androsterone and 5?-androstanediol) concentration in benign prostate tissue based on HSD3B1 genotype.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue gave two samples
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 15
Number analyzed (Tissue Sample) | 30
nM
  DHT homozygous(1245A): number analyzed (Participants) | 8
  DHT homozygous(1245A): number analyzed (Tissue Sample) | 16
  DHT homozygous(1245A) | 9.066 (7.775)
  T homozygous(1245A): number analyzed (Participants) | 8
  T homozygous(1245A): number analyzed (Tissue Sample) | 16
  T homozygous(1245A) | 6.901 (2.372)
  DHEA homozygous(1245A): number analyzed (Participants) | 8
  DHEA homozygous(1245A): number analyzed (Tissue Sample) | 16
  DHEA homozygous(1245A) | 46.110 (82.578)
  AD homozygous(1245A): number analyzed (Participants) | 8
  AD homozygous(1245A): number analyzed (Tissue Sample) | 16
  AD homozygous(1245A) | 8.394 (2.168)
  DHT heterozygous: number analyzed (Participants) | 5
  DHT heterozygous: number analyzed (Tissue Sample) | 10
  DHT heterozygous | 5.917 (3.458)
  T heterozygous: number analyzed (Participants) | 5
  T heterozygous: number analyzed (Tissue Sample) | 10
  T heterozygous | 4.929 (1.285)
  DHEA heterozygous: number analyzed (Participants) | 5
  DHEA heterozygous: number analyzed (Tissue Sample) | 10
  DHEA heterozygous | 18.5788 (13.02)
  AD heterozygous: number analyzed (Participants) | 5
  AD heterozygous: number analyzed (Tissue Sample) | 10
  AD heterozygous | 6.083 (2.5522)
  DHT homozygous (1245C): number analyzed (Participants) | 2
  DHT homozygous (1245C): number analyzed (Tissue Sample) | 4
  DHT homozygous (1245C) | 9.345 (5.607)
  T homozygous (1245C): number analyzed (Participants) | 2
  T homozygous (1245C): number analyzed (Tissue Sample) | 4
  T homozygous (1245C) | 4.704 (4.166)
  AD homozygous (1245C): number analyzed (Participants) | 2
  AD homozygous (1245C): number analyzed (Tissue Sample) | 4
  AD homozygous (1245C) | 8.303 (2.841)

3. Secondary Outcome: Other Androgens (DHT, T, DHEA, Androstenediol, 5α-dione, AD, Androsterone and 5α-androstanediol) Concentration in Malignant Prostate Tissue After Neo-adjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate the effect of neoadjuvant ARN-509 on other androgens (DHT, T, DHEA, androstenediol, 5?-dione, AD, androsterone and 5?-androstanediol) concentration in malignant prostate tissue after neoadjuvant leuprolide and ARN-509.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue gave two samples
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 24
Number analyzed (Tissue Sample) | 48
nM
  DHT homozygous (1245A): number analyzed (Participants) | 13
  DHT homozygous (1245A): number analyzed (Tissue Sample) | 26
  DHT homozygous (1245A) | 8.855 (7.4847)
  T homozygous (1245A): number analyzed (Participants) | 13
  T homozygous (1245A): number analyzed (Tissue Sample) | 26
  T homozygous (1245A) | 5.691 (2.531)
  DHEA homozygous (1245A): number analyzed (Participants) | 13
  DHEA homozygous (1245A): number analyzed (Tissue Sample) | 26
  DHEA homozygous (1245A) | 22.941 (11.523)
  AD homozygous (1245A): number analyzed (Participants) | 13
  AD homozygous (1245A): number analyzed (Tissue Sample) | 26
  AD homozygous (1245A) | 7.974 (4.005)
  DHT heterozygous: number analyzed (Participants) | 10
  DHT heterozygous: number analyzed (Tissue Sample) | 20
  DHT heterozygous | 5.238 (3.822)
  T heterozygous: number analyzed (Participants) | 10
  T heterozygous: number analyzed (Tissue Sample) | 20
  T heterozygous | 5.719 (3.513)
  DHEA heterozygous: number analyzed (Participants) | 10
  DHEA heterozygous: number analyzed (Tissue Sample) | 20
  DHEA heterozygous | 24.543 (16.779)
  AD heterozygous: number analyzed (Participants) | 10
  AD heterozygous: number analyzed (Tissue Sample) | 20
  AD heterozygous | 8.593 (3.736)
  DHT homozygous (1245C): number analyzed (Participants) | 1
  DHT homozygous (1245C): number analyzed (Tissue Sample) | 2
  DHT homozygous (1245C) | 2.622 (1.530)
  T homozygous (1245C): number analyzed (Participants) | 1
  T homozygous (1245C): number analyzed (Tissue Sample) | 2
  T homozygous (1245C) | 4.489 (1.197)
  DHEA homozygous (1245C): number analyzed (Participants) | 1
  DHEA homozygous (1245C): number analyzed (Tissue Sample) | 2
  DHEA homozygous (1245C) | 1.421 (0)
  AD homozygous (1245C): number analyzed (Participants) | 1
  AD homozygous (1245C): number analyzed (Tissue Sample) | 2
  AD homozygous (1245C) | 6.959 (3.956)

4. Secondary Outcome: To Compare the Level of DHT, T, DHEA, Androstenediol, 5alpha-dione, AD, Androsterone and 5alpha-androstanediol Between Normal and Malignant Prostate Tissue After Neoadjuvant Leuprolide and ARN-509.
Description: To compare the level of DHT, T, DHEA, androstenediol, 5alpha-dione, AD, androsterone and 5alpha-androstanediol between normal and malignant prostate tissue after neoadjuvant leuprolide and ARN-509.
Time Frame: Up to 28 Days
Population: Insufficent Tissue
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 54
Number analyzed (Tissue Sample) | 0

5. Secondary Outcome: PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C Expression (Via IHC) in Malignant Prostate Tissue After Neoadjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C tissue expression (via IHC) in malignant prostate tissue after treatment with Leuprolide and Apalutamide.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue for PSA and H3K27 were Analyzed. Two samples collected per participant. There was insufficient tissue for TMPRSS2, EZH2, H3K27, and UBE2C expression.
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 39
Number analyzed (Tissue Sample) | 78
nM
  PSA Homozygous (1245A): number analyzed (Participants) | 21
  PSA Homozygous (1245A): number analyzed (Tissue Sample) | 42
  PSA Homozygous (1245A) | 1.15 (0.662)
  H3K27 Homozygous (1245A): number analyzed (Participants) | 21
  H3K27 Homozygous (1245A): number analyzed (Tissue Sample) | 42
  H3K27 Homozygous (1245A) | 1.619 (0.882)
  PSA heterozygous: number analyzed (Participants) | 15
  PSA heterozygous: number analyzed (Tissue Sample) | 30
  PSA heterozygous | 1.393 (0.786)
  H3K27 heterozygous: number analyzed (Participants) | 15
  H3K27 heterozygous: number analyzed (Tissue Sample) | 30
  H3K27 heterozygous | 1.633 (0.890)
  PSA Homozygous (1245C): number analyzed (Participants) | 3
  PSA Homozygous (1245C): number analyzed (Tissue Sample) | 6
  PSA Homozygous (1245C) | 1.375 (1.500)
  H3K27 Homozygous (1245C): number analyzed (Participants) | 3
  H3K27 Homozygous (1245C): number analyzed (Tissue Sample) | 6
  H3K27 Homozygous (1245C) | 0.744 (0.756)

6. Secondary Outcome: PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C Expression (Via qPCR) in Malignant Prostate Tissue After Neoadjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C tissue expression (via qPCR) in malignant prostate tissue after treatment with Leuprolide and Apalutamide.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue for PSA, FKBP5, TMPRSS2 were analyzed. Two samples were collected from each participant. There was insufficient tissues for the EZH2, H3K27, and UBE2C expression.
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 39
Number analyzed (Tissue Sample) | 78
nM
  PSA homozygous (1245A): number analyzed (Participants) | 21
  PSA homozygous (1245A): number analyzed (Tissue Sample) | 42
  PSA homozygous (1245A) | 1.474 (1.488)
  FKBP5 homozygous (1245A): number analyzed (Participants) | 21
  FKBP5 homozygous (1245A): number analyzed (Tissue Sample) | 42
  FKBP5 homozygous (1245A) | 1.304 (0.874)
  TMPRSS2 homozygous (1245A): number analyzed (Participants) | 21
  TMPRSS2 homozygous (1245A): number analyzed (Tissue Sample) | 42
  TMPRSS2 homozygous (1245A) | 1.603 (1.071)
  PSA heterozygous: number analyzed (Participants) | 15
  PSA heterozygous: number analyzed (Tissue Sample) | 30
  PSA heterozygous | 1.127 (1.109)
  FKBP5 heterozygous: number analyzed (Participants) | 15
  FKBP5 heterozygous: number analyzed (Tissue Sample) | 30
  FKBP5 heterozygous | 1.127 (1.109)
  TMPRSS2 heterozygous: number analyzed (Participants) | 15
  TMPRSS2 heterozygous: number analyzed (Tissue Sample) | 30
  TMPRSS2 heterozygous | 1.742 (1.790)
  PSA homozygous (1245C): number analyzed (Participants) | 3
  PSA homozygous (1245C): number analyzed (Tissue Sample) | 6
  PSA homozygous (1245C) | 2.221 (1.027)
  FKBP5 homozygous (1245C): number analyzed (Participants) | 3
  FKBP5 homozygous (1245C): number analyzed (Tissue Sample) | 6
  FKBP5 homozygous (1245C) | 2.221 (1.027)
  TMPRSS2 homozygous (1245C): number analyzed (Participants) | 3
  TMPRSS2 homozygous (1245C): number analyzed (Tissue Sample) | 6
  TMPRSS2 homozygous (1245C) | 2.345 (1.145)

7. Secondary Outcome: PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C Expression (Via IHC) in Benign Prostate Tissue After Neoadjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate PSA, FKBP5, TMPRSS2, EZH2, H3K27 and UBE2C tissue expression (via IHC) in benign prostate tissue after treatment with Leuprolide and Apalutamide.
Time Frame: Up to 28 Days
Population: Insufficient tissue
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 54
Number analyzed (Tissue Sample) | 0

8. Secondary Outcome: PSA, FKBP5, TMPRSS2, EZH2, H3K27, and UBE2C Expression (Via qPCR) in Benign Prostate Tissue After Neoadjuvant Leuprolide and Apalutamide Based on Genotype Status.
Description: To evaluate PSA, FKBP5, TMPRSS2, EZH2, H3K27 and UBE2C tissue expression (via qPCR) in benign prostate tissue after treatment with Leuprolide and Apalutamide.
Time Frame: Up to 28 Days
Population: Insufficient Tissue
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 0

9. Primary Outcome: Dihydrotestosterone (DHT) Concentration in Malignant Prostate Tissue After a Combination Drug Treatment Based on Genotype Status
Description: To evaluate the differential effect of neo-adjuvant leuprolide and ARN-509 on dihydrotestosterone (DHT) concentration in malignant prostate tissue based on HSD3B1 genotype.
Time Frame: Up to 28 Days
Population: Participants with sufficient tissue each gave two samples
Measure: Mean (Standard Error); unit: nM
Units Other Than Participants: Tissue Sample
Arm/Group | Apalutamide + Leuprolide Acetate
Number analyzed (Participants) | 24
Number analyzed (Tissue Sample) | 48
nM
  homozygous (1245A): number analyzed (Participants) | 13
  homozygous (1245A): number analyzed (Tissue Sample) | 26
  homozygous (1245A) | 8.855 (7.4847)
  heterozygous (1254C): number analyzed (Participants) | 10
  heterozygous (1254C): number analyzed (Tissue Sample) | 20
  heterozygous (1254C) | 5.238 (3.822)
  homozygous (1245C): number analyzed (Participants) | 1
  homozygous (1245C): number analyzed (Tissue Sample) | 2
  homozygous (1245C) | 2.622 (1.530)

ADVERSE EVENTS:
Time Frame: Up to 8 Weeks following the last dose of study drug
Arm/Group | Apalutamide + Leuprolide Acetate
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 1/54
Other Adverse Events (participants affected / at risk) | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide + Leuprolide Acetate (N=54)
Genital Edema (Reproductive system and breast disorders) | 1 — Scrotal edema, discoloration, and hematuria expected post-operative changes, and not related to Apalutamide per investigator.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide + Leuprolide Acetate (N=54)
Anemia (Blood and lymphatic system disorders) | 3
Hypothyroidism (Endocrine disorders) | 9
Eye disorders - Other, specify (Intermittent dry & watering eyes) (Eye disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Edema, face (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 29
Localized edema (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Creatinine Increased (Investigations) | 4
Hyperglycemia (Investigations) | 5
Hyperkalemia (Investigations) | 4
Hypernatremia (Investigations) | 3
Hypoalbuminemia (Investigations) | 2
Hyponatremia (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 5
Platelet count decreased (Investigations) | 1
Weight Loss (Investigations) | 2
White blood cell decreased (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cognitive Disturbance (Nervous system disorders) | 3
Cognitive Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 9
Nervous system disorders - Other, specify (Restless leg syndrome (6); Mental fogginess (2)) (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 8
Libido decrease (Psychiatric disorders) | 3
Psychiatric disorders - Other, specify (Flat affect) (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 4
Urinary Retention (Renal and urinary disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Penis shrinkage) (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin disorder (2)) (Skin and subcutaneous tissue disorders) | 2
Hot Flashes (Vascular disorders) | 28
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02770391/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02770391/ICF_001.pdf